CLINICAL TRIAL: NCT00053378
Title: A Placebo-Controlled, Double-Blind Study to Examine the Use of Zemplar to Increase Serum Calcium Levels in ICU Subjects
Brief Title: A Study to Examine the Use of Zemplar to Increase Serum Calcium Levels in ICU Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: M01-395
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2006-08-02 (Estimated); Status verified 2006-07

CONDITIONS: Hypocalcemia
Keywords: hypocalcemia, ionized calcium, intensive care
MeSH Terms: conditions — Hypocalcemia | interventions — paricalcitol

INTERVENTIONS:
Drug: paricalcitol injection (Zemplar)
Behavioral: Effects on calcium regulation
Behavioral: Administration of elemental Ca during hypocalcemic ICU pts.

SUMMARY:
A study to determine the effect of Zemplar on the regulation of serum calcium levels and the need for administration of elemental calcium in hypocalcemic intensive care patients

ELIGIBILITY:
Inclusion Criteria:

* ICU patients APACHE III score between 70 - 150 at screening and within 24 hours of enrollment and a whole blood ionized calcium level less than 0.90 mmol/L or corrected whole blood calcium level less than or equal to 7.5 mg/dL.

Exclusion Criteria:

* Serum creatinine greater than 2.5 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2002-01

PRIMARY OUTCOMES:
The primary efficacy variable will be the change from Day 1 to last day of dosing in pH adjusted, serum ionized calcium levels.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Z Melnick, M.D., Study Director — Abbott
Locations (9):
- United States (9):
  - Merced Heart Association, Merced, California
  - Denver Health Medical Center, Denver, Colorado
  - Outcomes Research Institute, Hudson, Florida
  - Florida Hospital, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - Central Baptist Hospital Clinical Research Center, Lexington, Kentucky
  - Strong Memorial Hospital, Rochester, New York
  - St. Luke's Hospital, Bethlehem, Pennsylvania
  - Heart Care Associates, Hopewell, Virginia